CLINICAL TRIAL: NCT01570751
Title: A Trial Comparing the Efficacy, Patient-reported Outcomes and Safety of Insulin Degludec 200 U/mL vs Insulin Glargine in Subjects With Type 2 Diabetes Mellitus Requiring High-dose Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3943; U1111-1123-4774 (Other: WHO)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg followed by IGlar (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine
- IGlar followed by IDeg (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Cross-over trial, part 1: Individually adjusted IDeg administered subcutaneously (s.c., under the skin) once daily for 16 weeks in each treatment period.
Drug: insulin glargine — Cross-over trial, part 2: Individually adjusted IGlar administered subcutaneously (s.c., under the skin) once daily for the 16 week run-in period followed by 16 weeks in each treatment period.

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to confirm the efficacy of IDeg (insulin degludec) versus IGlar (insulin glargine) in controlling glycaemia. Subjects are to continue their pre-trial metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Current treatment with once daily insulin glargine in vials with a daily dose equal to or above 65 U and equal to or below 100 U
* Current treatment with a stable dose of metformin plus/minus one additional oral antidiabetic drug (OAD) for at least 12 weeks
* Glycosylated haemoglobin (HbA1c) equal to or above 7.5%

Exclusion Criteria:

* Current treatment with insulin other than insulin glargine in vials
* Treatment with thiazolidinediones or glucagon-like peptide-1 (GLP-1) receptor agonists within 12 weeks
* Stroke; heart failure; myocardial infarction; unstable angina pectoris; coronary arterial bypass graft or angioplasty
* Suffer from cancer (except basal cell skin cancer and squamous-cell cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (43):
- United States (42):
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Homestead, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Kingsville, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Schertz, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Novo Nordisk Investigational Site, Manatí, Puerto Rico

REFERENCES:
- [Result] Warren ML, Chaykin LB, Jabbour S, Sheikh-Ali M, Hansen CT, Nielsen TSS, Norwood P. Insulin Degludec 200 Units/mL Is Associated With Lower Injection Frequency and Improved Patient-Reported Outcomes Compared With Insulin Glargine 100 Units/mL in Patients With Type 2 Diabetes Requiring High-Dose Insulin. Clin Diabetes. 2017 Apr;35(2):90-95. doi: 10.2337/cd15-0058. PMID 28442823
- [Derived] Warren ML, Brod M, Hakan-Bloch J, Sparre T, Chaykin LB. Patient-reported outcomes from a randomized, crossover trial comparing a pen injector with insulin degludec versus a pen injector with insulin glargine U100 in patients with type 2 diabetes. Curr Med Res Opin. 2019 Sep;35(9):1623-1629. doi: 10.1080/03007995.2019.1605769. Epub 2019 May 21. PMID 30974973
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 37 sites in the United States of America (USA).
Pre-assignment Details: All subjects were on insulin glargine (IGlar, ≥ 65 U and ≤ 100 U/mL in 10 mL vials) treatment once daily (OD) administered subcutaneously at any time of day preferred by the subject for 16 week run-in period along with the daily pre-trial metformin dose.
Groups:
- IDeg/IGlar: The subjects in this arm for treatment period A received IDeg OD (200 U/mL in pre-filled pen device) subcutaneously (under the skin) for 16 weeks (treatment period A) followed by IGlar OD (100 U/mL in SoloStar® pen) for 16 weeks (treatment period B). Subjects were crossed over to IGlar without a wash-out period between the two treatment sequences. Subjects continued on metformin (pre-trial dose) throughout the trial. There was a follow-up visit 7 days following the last treatment visit.
- IGlar/IDeg: The subjects in this arm for treatment period A received IGlar OD (100 U/mL in SoloStar® pen) subcutaneously (under the skin) for 16 weeks (treatment period A) followed by IDeg OD (200 U/mL in pre-filled pen device) for 16 weeks (treatment period B). Subjects were crossed over to IDeg without a wash-out period between the two treatment sequences. Subjects continued on metformin (pre-trial dose) throughout the trial. There was a follow-up visit 7 days following the last treatment visit.
Period: Period A (16 Weeks)
Arm/Group | IDeg/IGlar | IGlar/IDeg
Started | 73 | 72
Exposed | 73 | 72
Completed | 70 | 67
Not Completed | 3 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal criteria | 0 | 1
Not completed — Unclassified | 2 | 3
Period: Period B (16 Weeks)
Arm/Group | IDeg/IGlar | IGlar/IDeg
Started | 70 | 67
Exposed | 70 | 67
Completed | 69 | 66
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: For 4 subjects baseline fasting plasma glucose (FPG) values were missing, hence did not contribute to the FPG summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg/IGlar | IGlar/IDeg | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.2) | 55.8 (9.0) | 55.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 42 | 48 | 90
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.0 (1.1) | 8.3 (1.4) | 8.2 (1.3)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 7.5 (3.3) | 8.5 (4.1) | 8.0 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 18) in Glycosylated Haemoglobin (HbA1c) at the End of Each 16 Week Treatment Period
Description: Values for change in HbA1c after each 16 weeks of treatment periods A and B.
Time Frame: Week 0, week 16 of each treatment period.
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). For 7 subjects in IDeg treatment A and 7 subjects in IGlar treatment B, HbA1c values were missing at the period of baseline and did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Groups:
- IDeg: Subjects received IDeg OD (200 U/mL in prefilled pen device) subcutaneously (under the skin) for 16 weeks in combination with metformin (pre-trial dose). As this was a 32-week cross-over trial with IGlar, subjects either received IDeg in treatment period A or treatment period B.
- IGlar: Subjects received IGlar OD (100 U/mL in Solostar® pen) subcutaneously (under the skin)for 16 weeks in combination with metformin (pre-trial dose). As this was a 32-week cross-over trial with IDeg, subjects either received IGlar in treatment period A or treatment period B.
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 138 | 138
percentage of glycosylated haemoglobin | -0.1 (1.1) | -0.1 (1.1)

2. Secondary Outcome: Change in Patient Reported Outcome (PRO) Scores From Baseline to the End of Each 16 Week Treatment Period
Description: Changes in subjects quality of life and insulin device satisfaction were evaluated using the following PROs: the Short-Form 36 Health Survey version 2 (SF-36) and the Treatment Related Impact Measure-Diabetes Device (TRIM-DD). PRO total scores were measured from baseline to the end of each 16-week treatment period. Responses were measured on a scale of 0 to 100, where higher scores indicated a better quality of life and higher insulin device satisfaction on the SF-36 and TRIM-DD questionnaires, respectively.
Time Frame: Week 0, week 16 of each treatment period.
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 8 subjects in each treatment group the values were missing at the period of baseline and did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 137 | 137
scores on a scale
  Physical score | -0.8 (7.7) | -0.6 (7.8)
  Mental score | 0.7 (9.3) | 0.4 (10.4)
  Total D-device | 11.0 (19.1) | 3.5 (19.1)

3. Secondary Outcome: Change in PRO Scores From the End of Treatment Period A Until After 4 Weeks of Treatment in Treatment Period B
Description: SF-36 and TRIM-DD total scores were measured at the end of treatment A (week 16) and 4 weeks into treatment B (week 20). Responses were measured on a scale of 0 to 100, where higher scores indicated a better quality of life and higher insulin device satisfaction on the SF-36 and TRIM-DD questionnaires, respectively.
Time Frame: Week 16, week 20
Population: The FAS included all randomised subjects. For 10 subjects, the PRO scores were missing.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IDeg/IGlar | IGlar/IDeg
Number analyzed (Participants) | 69 | 66
scores on a scale
  Physical score | 0.02 (7.07) | 0.60 (6.09)
  Mental score | 0.61 (8.88) | 0.21 (8.59)
  Total D-device | 10.24 (19.89) | -6.25 (11.10)

4. Secondary Outcome: Change From Baseline in Central Laboratory Measured Fasting Plasma Glucose (FPG) at the End of Each 16 Week Treatment Period
Description: Values of FPG in mmol/L from baseline to each 16 weeks of treatment periods.
Time Frame: Week 0, week 16, week 32
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 17 subjects in IDeg treatment A and 16 subjects in IGlar treatment B, FPG values were missing at the period of baseline and did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 128 | 129
mmol/L | -0.8 (4.2) | -0.0 (4.4)

5. Secondary Outcome: Change in FPG From the End of Treatment Period A Until After 4 Weeks of Treatment in Treatment Period B
Description: Values of FPG in mmol/L from the end of treatment period A until after 4 weeks of treatment in treatment period B.
Time Frame: Week 16, week 20
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 19 subjects the FPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg/IGlar | IGlar/IDeg
Number analyzed (Participants) | 63 | 63
mmol/L | -0.78 (3.41) | 0.19 (4.40)

6. Secondary Outcome: Number of Adverse Events (AEs)
Description: Number of treatment emergent adverse events (TEAEs) from week 0 to week 16 of the randomised treatment periods. A TEAE was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. TEAEs were attributed to the treatment given in the period in which the event occurred.
Time Frame: From baseline to the end of each 16 week treatment period.
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events
Arm/Group | IDeg | IGlar
Number analyzed (Participants) | 140 | 142
events | 105 | 111

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 32 weeks + 7 days follow up
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg | IGlar
Serious Adverse Events (participants affected / at risk) | 4/140 | 4/142
Other Adverse Events (participants affected / at risk) | 2/140 | 9/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=140) | IGlar (N=142)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=140) | IGlar (N=142)
Nasopharyngitis (Infections and infestations) | 2 (2) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.